CLINICAL TRIAL: NCT04677309
Title: Ultrasound Assessment of Aeration Changes After Lung Resection: a Pilot Study
Brief Title: LUS to Assess Lung Injury After Lung Resection
Acronym: THORUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ana Broseta Lleó (Other)
Collaborators: Hospital General Universitario de Valencia (Other)
Responsible Party: Sponsor-Investigator, Ana Broseta Lleó, Consultant in Anesthesiology, Hospital General Universitario de Valencia
Organization: Hospital General Universitario de Valencia (Other)
Other Study IDs: THORUS
Record Dates: First submitted 2020-11-24; First posted 2020-12-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Lung Neoplasm; Adult ALL; Lung Injury; Lung Injury, Ventilator Induced; Lung Inflammation; Lung Ischemia/Hypoxia; Postoperative Complications; Postoperative Respiratory Complication; Lung Cancer; Thoracic
Keywords: thoracic surgery; lung ultrasound; cytokines blood; lung injury; postoperative complications
MeSH Terms: conditions — Lung Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lung Injury; Ventilator-Induced Lung Injury; Pneumonia; Hypoxia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung resection less than lobectomy: participants scheduled for lung resection that is less than lobectomy
- Lung resection equal to or greater than lobectomy: participants scheduled for lung resection that is equal to or greater than lobectomy

SUMMARY:
The purpose of the study is to assess whether lung ultrasound is able to detect lung injury after lung resection surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are common after lung resection surgery, with an incidence that ranges between 11-32%. As PPC are associated with worse outcomes, many studies aim to find predictors that identify high risk patients and prompt specific interventions and/or monitoring and hence, improve outcomes. PPC result from lung injury inherent to lung resection surgery. Lung aeration changes seen with lung ultrasound (LUS) could detect lung injury and thus, identify patients at high risk of PPC. The underlying mechanisms of lung injury are different in the dependent and non-dependent lung; oxidative stress in both lungs, lung injury associated with one-lung ventilation in the dependent lung and ischemia/reperfusion or surgical manipulation in the non-dependent lung. LUS evaluates the operated and non-operated lung separately and so it can be valuable in understanding the characteristics and intensity of lung injury in each lung specifically.

This is a prospective, single-centre, observational study in which 28 consecutive participants with non-small cell lung cancer scheduled for lobectomy will be recruited. Participants will be divided in two groups depending on the surgical approach. First group will be lobectomy via thoracotomy. Second group will be lobectomy via VATS. Participants will be recruited consecutively until there are 14 patients in each group. LUS will be performed in each participant's dependent and non-dependent lung at three predefined time points: before surgery, after extubation and 24 h after surgery. Each hemithorax will be divided into 6 areas: anterior, lateral and posterior, separated by the anterior and posterior axillary lines, each divided into upper and lower zones. For each echographic examination, cineloops of the most pathological findings in each area will be stored and analysed offline by two independent and blinded anesthesiologists. From these, a semiquantitative score, the modified lung ultrasound score (mLUSS), will be calculated for each hemithorax to assess lung aeration at each time point. The level of agreement for mLUSS will be tested. At the same predefined time points blood plasma samples will be collected, flash-frozen and stored in order to measure levels of the inflammatory mediators IL-6, IL-10 and TNFα.

The invertigators hypothesise that LUS can detect lung injury after lung resection surgery. The primary objective of the study is to assess changes in lung aeration after lung resection with mLUSS. Secondary objectives are, first, to describe LUS findings after lung resection surgery, second, to assess the ability of mLUSS to detect oxygenation changes after lung resection and third, to compare the behaviour of inflammatory mediators in plasma with mLUSS changes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ASA I-III
* Non-small cell lung neoplasm
* Elective lung resection
* Via VATS
* Under one-lung ventilation

Exclusion Criteria:

* pregnancy
* Diagnosed pulmonary fibrosis
* Scheduled surgery limited to biopsy
* Surgery that includes resection of the thoracic wall or the diaphragm
* Predicted FEV1 < 40%
* Neoplasm metastasis
* Obesity class II or more (BMI ≥ 35 kg/m^2)
* Risk of malnutrition CONUT > 1
* Hemoglobin < 10 g/dl
* Chronic kidney failure: glomerular filtration < 60 ml/min/m^2, nephrectomy, kidney transplantation
* Treatment with corticosteroids or immunosuppressive agents 3 months before surgery
* Transfusion of blood products during the previous 10 days
* Heart failure (New York Heart Association Functional Class 3 or 4) during the week before surgery.
* Heart valve diseases over stage B of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines 2014
* Diastolic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients assigned to a tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in mLUSS after lung resection | preoperative vs immediate postoperative period vs 24 hours after surgery
  The modified lung ultrasound score (mLUSS) ranges 0-36; the higher the score, the less aeration (worse).

SECONDARY OUTCOMES:
LUS findings in the dependent and non-dependent lung | preoperative vs immediate postoperative period vs 24 hours after surgery
  description of LUS findings after lung resection surgery in each lung
Changes in oxygenation (PAFI) after lung resection | preoperative vs immediate postoperative vs 24 hours after surgery
  PAFI is the ratio between paO2 and fraction of inspired oxygen; the lower, the worse.
Changes in plasma cytokine IL-6 after lung resection | preoperative vs immediate postoperative vs 24 hours after surgery
Changes in plasma cytokine IL-10 after lung resection | preoperative vs immediate postoperative vs 24 hours after surgery
Changes in plasma TNFα after lung resection | preoperative vs immediate postoperative vs 24 hours after surgery
Changes in blood bone natriuretic peptide (BNP) after lung resection. | preoperative vs immediate postoperative vs 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ana Broseta Lleó, Consultant, Principal Investigator — Hospital General Universitario de Valencia
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No